CLINICAL TRIAL: NCT00729872
Title: A Phase 2a Randomized, Placebo-Controlled, Double-Blind, Multi-Center Dose Escalation Study, to Evaluate the Safety, Tolerability, Pharmacodynamics and Efficacy of AG011, in Subjects With Moderately Active Ulcerative Colitis
Brief Title: A Phase 2a Study to Evaluate the Safety, Tolerability, Pharmacodynamics and Efficacy of AG011 in Ulcerative Colitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ActoGeniX N.V. (Industry)
Responsible Party: Bernard Coulie, VP Research and Development, ActoGeniX
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG011-MDUC-201
Record Dates: First submitted 2008-08-04; First posted 2008-08-08 (Estimated); Last update posted 2009-09-10 (Estimated); Status verified 2009-09

CONDITIONS: Moderately Active Ulcerative Colitis
Keywords: AG011; Ulcerative Colitis; human Interleukin-10
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 (Experimental): AG011: low dose
  Interventions: Biological: AG011
- 2 (Placebo Comparator): Placebo: low dose
  Interventions: Other: Placebo
- 3 (Experimental): AG011: mid dose
  Interventions: Biological: AG011
- 4 (Placebo Comparator): Placebo: mid dose
  Interventions: Other: Placebo
- 5 (Experimental): AG011: high dose
  Interventions: Biological: AG011
- 6 (Placebo Comparator): Placebo: high dose
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AG011 — Capsules (low, mid or high dose), twice daily for 28 days, combined with Enema (low, mid or high dose respectively), once daily for 28 days.
  Arms: 1; 3; 5
Other: Placebo — Capsules (matching placebo for low, mid or high dose), twice daily for 28 days, combined with Enema (matching placebo for low, mid or high dose respectively), once daily for 28 days.
  Arms: 2; 4; 6

SUMMARY:
The purpose of this study is to verify the safety and tolerability of AG011 (genetically modified L. lactis that has been engineered to secrete human Interleukin-10), and to determine whether AG011 can successfully treat the symptoms of moderately active Ulcerative Colitis (UC).

DETAILED DESCRIPTION:
The purpose of this study is to verify the safety and tolerability of AG011 and to determine whether AG011 can successfully treat the symptoms of Ulcerative Colitis (UC). Three different dosages will be used in reference to a placebo.

AG011 is an experimental medication. It has been developed as potential treatment for moderately active UC.

AG011 is the clinical formulation of a genetically modified L. lactis that has been engineered to secrete human Interleukin-10 (hIL-10). By delivering hIL-10 locally at inflamed tissue in the intestine, it is believed that, compared to hIL-10 given by injection, the effectiveness may be increased, with fewer adverse effects.

Study medication will be provided in capsule and enema (topical rectal application) forms by ActoGeniX NV.

Subjects will be entered sequentially into one of three dose groups, starting from the lowest dose group. Within each of the first two dose groups, 15 subjects will be entered. Within the highest dose group, 30 subjects will be entered. Within each dose group, subjects will be randomly assigned in a 2:1 ratio to receive either AG011 or placebo for 28 days.

Timely monitoring of safety data is planned for the study, such that subject enrollment can continue without interruption for the purpose of data collection between dose groups. Safety and tolerability will be closely monitored by the Clinical Safety Specialist (CSS) assigned to the study. The CSS will review adverse events and laboratory safety data and report any safety concerns to the Sponsor and a Data Safety Monitoring Committee (DSMC).

At least 8 subjects must have safely completed study treatment for 28 days at a specific dose level, prior to escalation to the next dose group. The DSMC will convene to assess safety data when 8 subjects have completed study treatment for 28 days at the specific dose level. The role of the DSMC for the study will be complete when all subjects in the study have completed study treatment.

For those patients randomized within the active group, UC symptoms could improve. As a result of the information gathered by this study, the knowledge and understanding of UC could improve.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating females, 18 years of age or older. Females of child bearing potential must have negative serum or urine pregnancy tests at the screening visit and throughout the study, and must use a hormonal (oral, implantable or injectable) or barrier method of birth control throughout the study. Females unable to bear children must have documentation of such in the case report form (i.e. tubal ligation, hysterectomy, or post menopausal [defined as a minimum of one year since the last menstrual period]).
* Documented diagnosis of UC with a minimum disease extent of 15 cm from the anal verge.
* Presence of friability on endoscopy, with minimum of Grade 2 (modified Baron score) changes at approximately 15 cm or more from the anal verge.
* Minimum Mayo Clinic Disease Activity Score of 5, with a score of at least 1 on both the stool frequency and rectal bleeding components.
* Receiving 5-ASA treatment for at least two months and a stable dose of oral 5 ASA for at least two weeks prior to randomization. Concurrent treatment with prednisone, or equivalent glucocorticoid ≤ 20 mg/day is acceptable as follows: minimum dosing of 4 weeks prior to screening AND stable dose for 2 weeks prior to screening AND expected to remain on a constant dose during the trial. Use of 5-ASA compounds is not required for those subjects who have failed treatment with 5-ASA compounds, or are allergic or intolerant.
* Hepatic function (AST, ALT, total bilirubin, alkaline phosphatase, LDH) ≤ 2 times the upper limit of the normal range.
* Adequate renal function, as evidenced by serum creatinine ≤ 1.5 times the upper limit of the normal range.
* Hemoglobin ≥ 10 g/dL.
* ANC ≥ 1.5 x 10E9/L (1,500 mm3).
* Lymphocyte count ≥ 0.1 x 10E3/μL.
* Platelet count ≥ 100 x 10E9/L (100,000/mm3).
* Ability of subject to participate fully in all aspects of this clinical trial.
* Written informed consent must be obtained and documented.

Exclusion Criteria:

* Exhibiting severe ulcerative colitis as defined by the following criteria: ≥ 6 bloody stools daily with one or more of the following: oral temperature > 37.8 °C or > 100.0 °F, pulse > 90/min, hemoglobin < 10 g/dL.
* Crohn's disease.
* History of colectomy or partial colectomy.
* Clostridium (C.) difficile positive at screening visit or treated for C. difficile within the 4 weeks prior to randomization
* Treatment with antibiotics or probiotics at screening
* Treatment with cyclosporine, methotrexate, azathioprine, 6-MP, infliximab, adalimumab or other immunosuppressants/biologics within 4 weeks prior to randomization
* Use of rectal steroids or 5-ASA enemas within 2 weeks prior to randomization.
* Clinically significant active infection.
* Known chronic liver disease.
* Serious underlying disease other than UC in the opinion of the investigator.
* Alcohol or illicit drug consumption, which in the opinion of the investigator, may interfere with the subject's ability to comply with the study procedures
* Active psychiatric problems, which in the opinion of the investigator, may interfere with the subject's ability to comply with the study procedures.
* History of malignancy other than basal or squamous cell cancer of the skin that has been removed, or carcinoma in situ of the cervix that has been adequately treated.
* History of dysplasia in colonic biopsies.
* Receiving any investigational therapy or any approved therapy for investigational use within 30 days or 5 half-lives prior to randomization (whichever is longer).
* Pregnant or lactating women.
* Prior enrollment in the current study and had received study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
SAFETY: Adverse Events | day 1, 8 15, 22, 29, 57
SAFETY: Physical Examination (complete or brief) | day -7, 1, 8, 15, 22, 29
SAFETY: Vital signs | day -7, 1, 8, 15, 22, 29, 57
SAFETY: Clinical Laboratory Tests (hematology, serum chemistry, urinalysis) | day -7, 1, 8, 15, 22, 29, 57
SAFETY: Analysis of hIL-10 (systemic exposure) and anti-hIL-10 antibodies (immunogenicity) in plasma | day 1, day 29
SAFETY: Stool Diary | From day -7 until day 29
SAFETY: Other Safety Measures (Stool samples for culture, ova and parasite evaluation and Clostridium difficile assay. | day -7
BIOLOGICAL CONTAINMENT: Evaluation of living, genetically modified micro-organisms in stool samples | day 1, 8, 36
PHARMACODYNAMICS: Biomarkers in blood and colon biopsy samples | day -7, 29

SECONDARY OUTCOMES:
EFFICACY: Flexible sigmoidoscopy (assessment of inflammation) | Day -7, 29
EFFICACY: Histological assessment of inflammation (biopsy samples) | Day -7, 29
EFFICACY: Disease activity assessments (MCDAS, UCCS, Investigator and Subject Global Ratings) | Day -7, 1, 8, 15, 22, 29, 57
EFFICACY: Laboratory assessments (CRP and fecal calprotectin) | Day 1, 15, 29, 57

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Coulie, MD PhD, Study Chair — Chief Medical Officer ActoGeniX NV; Annegret Van der Aa, PhD, Study Director — Project Manager ActoGeniX NV; Severine Vermeire, MD PhD, Principal Investigator — UZ Leuven, Belgium; Geert D'Haens, MD PhD, Principal Investigator — Imelda Bonheiden, Belgium; Martine De Vos, MD PhD, Principal Investigator — UZ Gent, Belgium; Tom Moreels, MD PhD, Principal Investigator — UZ Antwerpen, Belgium; Daan Hommes, MD PhD, Principal Investigator — Leiden University Medical Center; Erik Hertervig, MD PhD, Principal Investigator — Lund University Hospital, Sweden; Curt Tysk, MD PhD, Principal Investigator — Orebro University Hospital, Sweden; Robert Lofberg, MD PhD, Principal Investigator — Karolinska Institutet; Pierre Paré, MD PhD, Principal Investigator — Hôpital St-Sacrement Quebec, Canada; William Barnett, MD PhD, Principal Investigator — LHSC - University Campus London, Canada; Brian Bressler, MD PhD, Principal Investigator — GI Research Institute Vancouver, Canada; James Gregor, MD PhD, Principal Investigator — LHSC - South Street Campus London, Canada; Hillary Steinhart, MD PhD, Principal Investigator — Mount Sinai Hospital, Canada; Richmond Sy, MD PhD, Principal Investigator — Ottawa Hospital General Campus, Canada; William Depew, MD PhD, Principal Investigator — Hotel-Dieu Hospital Kingston, Canada; Donald Daly, MD PhD, Principal Investigator — Victoria BC, Canada; Philippe Vergauwe, MD PhD, Principal Investigator — AZ Groeninge Campus St.-Niklaas Kortrijk, Belgium; Olivier Dewit, MD PhD, Principal Investigator — UCL St. Luc Brussels, Belgium
Locations (18):
- Belgium (6):
  - Imelda Bonheiden, Bonheiden
  - UCL St. Luc, Brussels
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
  - AZ Groeninge Campus St.-Niklaas, Kortrijk
  - UZ Leuven, Leuven
- Canada (8):
  - GI Research Institute, Vancouver, British Columbia
  - The office of Dr. Donald Daly, Victoria, British Columbia
  - Hotel Dieu Hospital, Kingston, Ontario
  - LHSC - South Street Campus, London, Ontario
  - LHSC - University Campus, London, Ontario
  - Ottawa Hospital General Campus, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Hôpital St-Sacrement, Québec, Quebec
- Leiden University Medical Center, Leiden, Netherlands
- Sweden (3):
  - Lund University Hospital, Lund
  - Orebro University Hospital, Örebro
  - Sophiahemmet, Stockholm

REFERENCES:
- [Background] Braat H, Rottiers P, Hommes DW, Huyghebaert N, Remaut E, Remon JP, van Deventer SJ, Neirynck S, Peppelenbosch MP, Steidler L. A phase I trial with transgenic bacteria expressing interleukin-10 in Crohn's disease. Clin Gastroenterol Hepatol. 2006 Jun;4(6):754-9. doi: 10.1016/j.cgh.2006.03.028. Epub 2006 May 22. PMID 16716759
- [Derived] Robert S, Steidler L. Recombinant Lactococcus lactis can make the difference in antigen-specific immune tolerance induction, the Type 1 Diabetes case. Microb Cell Fact. 2014 Aug 29;13 Suppl 1(Suppl 1):S11. doi: 10.1186/1475-2859-13-S1-S11. Epub 2014 Aug 29. PMID 25185797